CLINICAL TRIAL: NCT03665155
Title: First-in- Human Imaging of Multiple Myeloma Using 89Zr-DFO-daratumumab, a CD38-targeting Monoclonal Antibody
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-267
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: 89Zr-DFO-daratumumab; CD38-targeting monoclonal antibody; CT; MR; FDG PET/CT; 18-267
MeSH Terms: conditions — Multiple Myeloma | interventions — Positron Emission Tomography Computed Tomography; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a phase I/II study with the goal to assess the feasibility of using the anti-CD38 monoclonal antibody daratumumab, labeled with Zirconium-89 (89Zr ) through deferoxamine (DFO), known as 89Zr-DFO-daratumumab, for PET imaging of multiple myeloma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-daratumumab (Experimental): Three patients will be administered 2 mCi of 89Zr-daratumumab in a total of 50 mg of daratumumab antibody. Administered activity (1 to 5 mCi) of radioactivity and total amount of administered antibody (3 to 50 mg) will be adjusted in subsequent patients in order to maximize image quality.
  Patients in phase I will have up to 4 PET/CT scans, multiple blood draws, whole-body counts, and safety monitoring to determine pharmacokinetics, radiation dosimetry, and safety of 89Zr-DFO-daratumumab for PET/CT imaging. Phase II (total of 21-24 patients). After pharmacokinetics and radiation dosimetry are determined in phase I, additional patients will be enrolled in phase II.
  Interventions: Drug: 89Zr-daratumumab; Device: PET/CT scans; Other: Blood draws

INTERVENTIONS:
Drug: 89Zr-daratumumab — 2 mCi of 89Zr-daratumumab will be administered on day 0.
Device: PET/CT scans — PET/CT images will be obtained on post-administration days 1, 2-4, 5-6, and/or 7-8 following administration of 89Zr-DFO-daratumumab to determine the optimal time point for imaging.
Other: Blood draws — Blood and serum samples will be weighed and counted in a scintillation well counter calibrated for 89Zr. Immediately before or after each PET/CT imaging session,

SUMMARY:
The purpose of this study is to test 89Zr-DFO-daratumumab, a new imaging agent, to demonstrate its safety and ability to take pictures of the myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or greater
* Histologically/Immunohistochemistry confirmed CD38-positive multiple myeloma
* At least one tumor lesion on CT, MRI, or FDG PET/CT within 60 days of protocol enrollment
* ECOG performance status 0 to 2
* For Phase II patients only: plan for initiation of standard-of-care daratumumab/lenalidomide therapy.

Exclusion Criteria:

* Life expectancy < 3 months
* Pregnancy or lactation
* Patients who cannot undergo PET/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 450 pounds.
* History of anaphylactic reaction to humanized or human antibodies or a Grade 3 or 4 administration reaction during a daratumumab administration.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ulaner, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Slaon-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase I portion of the study has concluded. The Phase II portion will not open due to the study PI leaving the institution.
Groups:
- Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody: Phase I: Dose Escalation 1-5 mCi in 50mg of antibody
- Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody: Phase I: Dose Escalation 1-5 mCi in 20mg of antibody
- Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody: Phase I: Dose Escalation 1-5 mCi in 3-50mg of antibody
Period: Overall Study
Arm/Group | Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody | Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody | Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody
Started | 3 | 7 | 1
Completed | 3 | 7 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody | Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody | Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody | Total
Number analyzed (Participants) | 3 | 7 | 1 | 11
Age, Continuous [Mean (Full Range); unit: years] | 60 [54 to 70] | 58.4 [37 to 80] | 60 [60 to 60] | 59 [37 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 2 | 5 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 1 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 5 | 0 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 7 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Average Absorbed Radiation Dose Estimates for Normal Tissues for Phase I Participants
Description: Standardized uptake value (SUV) in various organs will be estimated from VOI analysis of clinical images and converted to activity-time curves. The areas under the activity-time curves will be derived by integration, converted to residence times, and used as input to the OLINDA/EXM dosimetry program to obtain absorbed dose estimates for normal tissues for all Phase I participants, regardless of study dose. Each participant underwent four PET/CT scans over the next 8 days, as well as blood chemistry and whole-body counts, to determine safety, tracer biodistribution, pharmacokinetics, and radiation dosimetry. Because 89Zr has a half-life of 78 hours, only a single administration of tracer was needed to obtain all four PET/CT scans for all Phase I participants. Results were combined because all received the same dose of tracer.
Time Frame: up to 19 months
Measure: Mean (Standard Error); unit: mSv/MBq
Groups:
- 89Zr-daratumumab: The Phase I portion of the study has concluded. The Phase II portion has not yet opened to accrual.
Arm/Group | 89Zr-daratumumab
Number analyzed (Participants) | 11
mSv/MBq | 0.49 (0.07)

ADVERSE EVENTS:
Time Frame: approximately 1 year 7 months
Groups:
- Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody; Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody; Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody: Three patients will be administered 2 mCi of 89Zr-daratumumab in a total of 50 mg of daratumumab antibody. Administered activity (1 to 5 mCi) of radioactivity and total amount of administered antibody (3 to 50 mg) will be adjusted in subsequent patients in order to maximize image quality.
  Patients in phase I will have up to 4 PET/CT scans, multiple blood draws, whole-body counts, and safety monitoring to determine pharmacokinetics, radiation dosimetry, and safety of 89Zr-DFO-daratumumab for PET/CT imaging. Phase II (total of 21-24 patients).
Arm/Group | Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody | Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody | Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 5/7 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody (N=3) | Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody (N=7) | Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody (N=1)
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Escalation 1-5 mCi in 50mg of Antibody (N=3) | Phase I: Dose Escalation 1-5 mCi in 20mg of Antibody (N=7) | Phase I: Dose Escalation 1-5 mCi in 3-50mg of Antibody (N=1)
Lymphocyte count decreased (Investigations) | 2 | 4 | 0
Neutrophil count decreased (Investigations) | 2 | 2 | 0
White blood cell decreased (Investigations) | 2 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT03665155/Prot_SAP_000.pdf